CLINICAL TRIAL: NCT04746911
Title: An Open Label, 4-Week, Phase 2, Maximal Usage Pharmacokinetics and Safety Study of ARQ-151 Cream 0.3% Administered QD in Pediatric Subjects (Ages 2 to 5 Years Old) With Plaque Psoriasis
Brief Title: Maximal Usage Pharmacokinetics and Safety of ARQ-151 in Children With Plaque Psoriasis (ARQ-151-216)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-216
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 cream 0.3% (Experimental): Open label study of ARQ-151 cream 0.3% applied once daily for 4 weeks
  Interventions: Drug: ARQ-151 cream 0.3%

INTERVENTIONS:
Drug: ARQ-151 cream 0.3% — ARQ-151 cream 0.3% applied to chronic plaque psoriasis lesions once a day for 4 weeks
  Other Names: Topical roflumilast

SUMMARY:
This is a Phase 2, open label, maximal usage PK and safety study of ARQ-151 cream 0.3% in pediatric subjects (ages 2 to 5 years old) with plaque psoriasis:

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent(s) or legal guardian.
* Males or females, 2 to 5 years old (inclusive).
* Clinical diagnosis of psoriasis vulgaris of at least 2 months duration as determined by the Investigator or through subject interview. Stable disease for the past 3 weeks.
* Psoriasis vulgaris on the face, extremities, trunk, and/or intertriginous areas involving at least 2% of BSA (excluding the scalp, palms, and soles).
* An Investigator Global Assessment of disease severity (IGA) of at least Mild ('2') at Baseline.
* Subject has adequate venous access for PK sampling in areas not involved by plaque psoriasis and not being treated with ARQ-151 (e.g., back of the hands).
* In good health as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry labs and hematology values.
* Subjects and parent(s)/legal guardian(s) are considered reliable and capable of adhering to the Protocol and Visit Schedule, according to the judgment of the Investigator.

Exclusion Criteria:

* Subjects with any serious medical or psychiatric condition or clinically significant laboratory, ECG, vital signs, or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.
* Planned initiation or changes to concomitant medication that could, in the opinion of the Investigator, affect psoriasis vulgaris
* Current diagnosis of non-plaque form of psoriasis (e.g., guttate, erythrodermic/exfoliative, palmoplantar only involvement, or pustular psoriasis). Current diagnosis of drug-induced psoriasis.
* Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
* Subjects who cannot discontinue the use of strong cytochrome P-450 CYP3A4 inducers for 2 weeks prior to Baseline/Day 1and during the study period.
* Subjects who cannot discontinue the use of strong cytochrome P-450 CYP3A4 inhibitors for 2 weeks prior to Baseline/Day 1 and during the study period.
* Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Day 1 and during the study.
* Subjects who cannot discontinue specific systemic therapies and/or topical therapies prior to the Baseline/Day 1 and during the study period according to the protocol.
* Subjects with any infection requiring oral or intravenous administration of antibiotics, antifungal or antiviral agents within 2 weeks prior to Baseline/Day 1.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) profile of ARQ-151 cream 0.3% and its major N-oxide metabolite | Week 4
  Plasma levels of circulating roflumilast and its major N-oxide metabolite
Incidence of adverse events | Week 4
  Number of participants with adverse events during treatment will be assessed
Incidence of application site reactions | Week 4
  Number of subjects that experience an application site skin reaction by investigator assessment and application site reactions reported as adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (18):
- United States (16):
  - Arcutis Clinical Site 603, Mountain Brook, Alabama
  - Arcutis Clinical Site 604, Scottsdale, Arizona
  - Arcutis Clinical Site 609, Fountain Valley, California
  - Arcutis Clinical Site 618, Los Angeles, California
  - Arcutis Clinical Site 608, Los Angeles, California
  - Arcutis Clinical Site 611, Rancho Santa Margarita, California
  - Arcutis Clinical Site 610, Boca Raton, Florida
  - Arcutis Clinical Site 602, Coral Gables, Florida
  - Arcutis Clinical Site 613, Delray Beach, Florida
  - Arcutis Clinical Study Site 628, Miami, Florida
  - Arcutis Clinical Site 607, Miami, Florida
  - Arcutis Clinical Site 627, West Lafayette, Indiana
  - Arcutis Clinical Site 606, Arlington, Texas
  - Arcutis Clinical Site 619, Frisco, Texas
  - Arcutis Clinical Study Site 619, Frisco, Texas
  - Arcutis Clinical Site 605, Houston, Texas
- Arcutis Clinical Site 621, Toronto, Ontario, Canada
- Arcutis Clinical Site 630, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Hebert AA, Guide SV, Groysman V, Gonzalez ME, Blanco D, Laquer V, Seal MS, Thurston A, Krupa D, Snyder S, Burnett P, Chu DH, Berk DR, Higham RC. Early Evidence of Safety, Clinical Benefit, and Pharmacokinetics of Roflumilast Cream 0.3% Once Daily for Treatment of Mild or Moderate Plaque Psoriasis in Children Aged 2-11 Years. Pediatr Dermatol. 2026 Jan-Feb;43(1):105-108. doi: 10.1111/pde.70013. Epub 2025 Aug 27. PMID 40862624